CLINICAL TRIAL: NCT06304662
Title: Physical and Mental Health. Effects of Yoga as a Therapeutic Tool.
Brief Title: Yoga for Physical and Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: *University of Jaén
Record Dates: First submitted 2024-03-03; First posted 2024-03-12 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group (CG) that is not going to undergo treatment, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity, and they will be given the guide of recommendations for the promotion of physical activity.
- Experimental Group (Experimental): The experimental group (EG) that after an initial evaluation will be subjected to a physical training program based on the ERFS, for 12 weeks with 3 weekly sessions (Monday, Wednesday and Friday), with a duration of 30-45 min per session. Once the intervention is finished, a final evaluation will be used again to see if there is a difference or not with the results obtained at the beginning.
  Interventions: Other: Yoga intervention

INTERVENTIONS:
Other: Yoga intervention — Over 12 weeks, students will attend 50-minute yoga sessions twice a week. Sessions start with 10 minutes of mindful breathing and gentle warm-up movements, followed by 30 minutes of tailored yoga postures for relaxation and stretching. Students progress from basic to advanced postures, with adaptations for individual needs. Each session ends with a guided meditation for inner calm. A 10-minute cool-down encourages deep relaxation. Emphasis is on stress reduction, flexibility, and mindfulness, tailored to university life challenges. Continuous assessment ensures sessions meet students' evolving needs and optimize yoga's benefits in the university setting.
  Arms: Experimental Group

SUMMARY:
In the university environment, where academic pressure and personal exploration are paramount, yoga serves as a sanctuary for students facing stress and seeking self-discovery. Through practices like asanas, pranayama, and meditation, yoga equips students with tools to manage stress, foster inner balance, and enhance emotional well-being. Apart from its emotional benefits, yoga offers physical advantages, improving strength, flexibility, and posture, particularly beneficial for those sedentary due to academic demands. Moreover, yoga enhances concentration and mental clarity through mindfulness practices, aiding students in academic focus and problem-solving.Additionally, yoga provides a space for students to disconnect from external stimuli and recharge, reducing mental and physical fatigue while boosting vitality. By integrating yoga into university life, students can better balance academic pressures with personal care, laying the groundwork for a more harmonious and mindful future.

ELIGIBILITY:
Inclusion Criteria:

* University students who do not participate in any physical exercise program
* Sufficient physical autonomy to participate in the physical activities required by the study
* That they are able to understand the instructions, programs and protocols of this project.

Exclusion Criteria:- University students who have serious physical or mental conditions

* Lack of commitment to regular attendance
* Extensive previous experience in yoga

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Stress level | Up to twelve weeks
  Perceived Stress Scale (PSS). This scale is a self-report instrument that evaluates the level of perceived stress during the last month, it consists of 14 items with a response format of a five-point scale (0 = never, 1 = almost never, 2 = occasionally when, 3 = often, 4 = very often). The total score of the PSS is obtained by reversing the scores of items 4, 5, 6, 7, 9, 10 and 13 (in the following sense: 0=4, 1=3, 2=2, 3=1 and 4 =0) and then adding the 14 items. The direct score obtained indicates that a higher score corresponds to a higher level of perceived stress.

SECONDARY OUTCOMES:
D2 test | Up to twelve weeks
  Evaluates selective attention and concentration in the school context. The participant's task is to check carefully, starting from left to right, what is written on each line and must mark all the letters that have two small lines (two below, two above or one below and one above) with a "d". ". These elements are considered relevant. The other combinations (the "d" and the "p", with and without dashes) are considered irrelevant and should not be marked. The participant has 20 s for each line. This test has shown excellent reliability, with ranges between 0.90 and 0.97 for both Cronbach's α and the test-retest, and has also shown convergent and divergent validity.
Mindful Attention Awareness Scale (MAAS) | Up to twelve weeks
  It evaluates, in a global way, the dispositional capacity of an individual to be attentive and aware of the experience of the present moment in everyday life. The scale is a 15-item univariate self-report with a view of the mindfulness construct centered on the attention / consciousness variable.
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess hand grip strength.
Anxiety and Depression | Up to twelve weeks
  Hospital Anxiety and Depression Scale (HADS). This scale consists of 14 items with 4 response alternatives ranging from 0 to 3 for a total of 0 to 21 points. It has 2 subscales and the score is obtained by adding the scores of each item that make it up, the interpretation criteria being the following: Range of normality (0-7), Possible case of anxiety or depression (8-10) and Case of anxiety or depression (11-21).
Sleep quality | Up to twelve weeks
  Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of 19 self-assessment questions or items and 5 more to be completed by the person with whom the participant shares a bed or room (although the latter is only used to provide clinical information). These items generate a total score and 7 components or domains: sleep quality; sleep latency; sleep duration; sleep efficiency; sleep disorders; use of sleeping medications; daytime dysfunction. The PSQI total score ranges from 0 to 21, with a higher score indicating poorer sleep quality.
The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | Up to twelve weeks
  is a 14-items questionnaire of mental well-being including subjective well-being and psychological functioning. All items in a 5-point Likert scale are worded positively and addressed aspects of positive mental health and measure the frequency of the subject's attitudes from "never" to "always". Higher scores indicate mental well-being. The Italian version of the WEMWB proved to be a reliable instrument, as indicated by a Cronbach's alpha that ranged from 0.83 to 0.864. The authors of the Italian WEMWBS reported for the students a mean score of 41.45 ± 6.66.
Difficulties in Emotion Regulation Scale (DERS) | Up to twelve weeks
  It is one of the most used tests to evaluate emotional control problems in adults. The 36-item self-report scale is used to generate scores on the following six subscales by asking respondents how they connect with their emotions: a) non-acceptance of emotional responses; b) difficulty engaging in goal-directed behavior; c) difficulties in impulse control; d) lack of emotional awareness; e) Limited access to emotion regulation strategies; and f) lack of emotional clarity. To rate each item, a 5-point Likert scale is used, from 1 which is "almost never" to 5 which is "almost always". A higher score indicates greater difficulties in regulating emotions, in other words, greater emotional dysregulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No